CLINICAL TRIAL: NCT02216331
Title: A Phase I Open-label Trial to Investigate the Pharmacokinetic Interaction Between Rifapentine or Rifampicin and a Single Dose of TMC207 in Healthy Subjects
Brief Title: PK Interaction Between Rifapentine or Rifampicin and a Single Dose of TMC207 in Healthy Subjects (TMC207-CL002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC207-CL002
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; PK; TMC207; bedaquiline; rifapentine; rifampicin; drug drug interaction
MeSH Terms: conditions — Tuberculosis | interventions — bedaquiline; rifapentine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 TMC207 alone (Experimental): A single 400 mg dose of TMC207 will be administered as 4 tablets of 100 mg per tablet on Study Day 1.
  Interventions: Drug: TMC207
- Group 1 TMC207 and rifapentine (Experimental): A single 400 mg dose of TMC207 will be administered as 4 tablets of 100 mg per tablet on Study Day 29 and 600 mg of rifapentine administered as 4 tablets of 150 mg per tablet on each of Study Days 20-41.
  Interventions: Drug: TMC207; Drug: rifapentine
- Group 2 TMC207 alone (Experimental): A single 400 mg dose of TMC207 will be administered as 4 tablets of 100 mg per tablet on Study Day 1.
  Interventions: Drug: TMC207
- Group 2 TMC207 and rifampicin (Experimental): A single 400 mg dose of TMC207 will be administered as 4 tablets of 100 mg per tablet on Study Day 29 and 600 mg of rifampicin administered as 4 capsules of 150 mg per capsule on each of Study Days 20-41.
  Interventions: Drug: TMC207; Drug: rifampicin

INTERVENTIONS:
Drug: TMC207 — This is a two group, 2 period study design with both groups in the first period receiving TMC207 alone, followed by one group in the second period receiving TMC207 in the presence of dosing with rifapentine and the other group receiving TMC207 in the presence of dosing with rifampicin. All treatments details specified under "Arms" description.
  Other Names: bedaquiline
Drug: rifapentine
  Arms: Group 1 TMC207 and rifapentine
Drug: rifampicin
  Arms: Group 2 TMC207 and rifampicin

SUMMARY:
This is a open-label study, 2-treatment, 2-period, single sequence design. Period 1 will examine the pharmacokinetics of TMC207 in the absence of rifapentine or rifampicin. Subjects will receive a single 400-mg dose of TMC207 administered alone on Study Day 1. Period 2 will examine the effects of repeated doses of either rifapentine or rifampicin on TMC207 pharmacokinetics and will begin on Study Day 20. During Period 2, subjects will receive 22 daily doses of either 600 mg rifapentine or rifampicin from Study Day 20 through Study Day 41. A single 400-mg dose of TMC207 will be administered on Study Day 29. Subjects will be confined to the clinic from Study Day-1 to Study Day 2 in the morning of Period 1, and Study Day 19 to Study Day 30 in the morning of Period 2. The study hypothesis is to determine whether Rifapentine affects the pharmacokinetics of TMC207 as measured by effects on Cmax and AUC(0-t) to a lesser degree than rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 55 years, extremes included.
* Non tobacco/nicotine using (at least 3 months prior to screening).
* Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 32.0 kg/m2, inclusive.
* Informed Consent Form (ICF) signed voluntarily before the first trial-related activity.
* Able to comply with protocol requirements.
* Healthy on the basis of a medical evaluation or history that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, and hematology tests and a urinalysis carried out at screening (See Section 6.1).

Exclusion Criteria:

* Female, except if postmenopausal since more than 2 years, or post-hysterectomy, or post surgical sterilization, i.e., tubal ligation (without reversal operation) or total hysterectomy.
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures.
* Any clinically significant (as deemed by the Principle Investigator) history acute illness (resolved within 4 weeks of screening), or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic, psychological, or psychiatric disease.
* Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability.
* Any history of significant skin disease such as, but not limited to, rash or eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria. Subjects with a history of skin disease may be enrolled into the study after consultation with the Sponsor Medical Monitor.
* Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial (i.e. rifapentine, rifampicin, and TMC207).
* Subjects with QTcF [Fredericia correction] interval > 450 msec (based on the average of the triplicate ECGs) at screening (and confirmed by repeat ECG).
* Subjects with any other clinically significant ECG abnormality at screening, such as arrhythmia, ischemia, or evidence of heart failure or with a family history of Long QT Syndrome.
* Use of concomitant medication, including over-the-counter products and dietary supplements, except for ibuprofen and paracetamol up to 7 days before the first dose of trial medication and all prescribed medication must have been discontinued at least 14 days before first intake of trial medication.
* Participation in an investigational drug trial within 60 days prior to the first intake of trial medication.
* Donation of blood or significant loss of blood within 56 days or plasma donation within 7 days preceding the first intake of trial medication.
* Having received TMC207 in a previous trial.
* Positive HIV-1 or HIV-2 test at screening
* Hepatitis A, B, or C infection (confirmed by hepatitis A antibody IgM, hepatitis B surface antigen, or hepatitis C virus antibody, respectively) at screening.
* A positive urine drug test at screening. Urine will be tested to check the current use of alcohol, amphetamines, benzodiazepines, cocaine, cannabinoids, and opioids.
* Subjects with the following laboratory abnormalities at screening as defined by the NIH, NIAID, Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table and in accordance with the normal ranges of the clinical laboratory: Serum creatinine grade 1 or greater (> 1.0 x ULN); Pancreatic lipase grade 1 or greater (> 1.0 x ULN); Hemoglobin grade 1 or greater (≤ 10.5 g/dL); Platelet count grade 1 or greater (≤ 99000/mm3); Absolute neutrophil count grade 1 or greater (≤ 1500/mm3); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (> 1.0 x ULN); Total bilirubin grade 1 or greater (> 1.0 x ULN); Any other toxicity grade 2 or above, including: proteinuria (spot urine) > 1+ and gross hematuria.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed TMC207 concentration in ng/mL [Cmax] between Groups 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on Cmax of TMC207, the Cmax of TMC207 was compared between Group 1 (rifapentine) and Group 2 (rifampicin) using analysis of variance model (ANOVA).
Area under the TMC207 concentration-time curve in ng*hr/mL [AUC0-t] between Groups 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on AUC0-t of TMC207, the AUC0-t of TMC207 was compared between Group 1 (rifapentine) and Group 2 (rifampicin) using analysis of variance model (ANOVA).
Area under the TMC207 concentration cuve from time zero to infinity in ng*hr/mL [AUC0-inf] between Groups 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on AUC0-inf of TMC207, the AUC0-inf of TMC207 was compared between Group 1 (rifapentine) and Group 2 (rifampicin) using analysis of variance model (ANOVA).

SECONDARY OUTCOMES:
Maximum observed TMC207 concentration in ng/mL [Cmax] within treatment groups between Periods 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on Cmax of TMC207, the Cmax of TMC207 was compared between the TMC207 + rifapentine treatment (Group 1) or rifampicin (Group 2) and TMC207 alone using analysis of variance model (ANOVA).
Area under the TMC207 concentration-time curve in ng*hr/mL [AUC0-t] within treatment groups between Periods 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on AUC0-t of TMC207, the AUC0-t of TMC207 was compared between the TMC207 + rifapentine treatment (Group 1) or rifampicin (Group 2) and TMC207 alone using analysis of variance model (ANOVA).
Area under the TMC207 concentration cuve from time zero to infinity in ng*hr/mL [AUC0-inf] within treatment groups between Periods 1 and 2 | through 336 hours post dosing in Period 1 and Period 2
  To evaluate the relative effect of rifapentine and rifampicin on AUC0-inf of TMC207, the AUC0-inf of TMC207 was compared between the TMC207 + rifapentine treatment (Group 1) or rifampicin (Group 2) and TMC207 alone using analysis of variance model (ANOVA).

OTHER OUTCOMES:
Number of participants with adverse events | through study day 57
  To compare the safety and tolerability as measured by the number of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion (MDS Pharma Services)
Locations (1):
- Celerion (MDS Pharma Services), Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Winter H, Egizi E, Murray S, Erondu N, Ginsberg A, Rouse DJ, Severynse-Stevens D, Pauli E. Evaluation of the pharmacokinetic interaction between repeated doses of rifapentine or rifampin and a single dose of bedaquiline in healthy adult subjects. Antimicrob Agents Chemother. 2015 Feb;59(2):1219-24. doi: 10.1128/AAC.04171-14. Epub 2014 Dec 15. PMID 25512422
- See also: Global Alliance for TB Drug Development website — http://www.tballiance.org